CLINICAL TRIAL: NCT05826444
Title: Morphological and Functional Phenotype of Isolated Microvascular Cardiac Allograft Vasculopathy in Heart Transplant Recipients
Brief Title: Microvascular Cardiac Allograft Vasculopathy Trial
Acronym: mCAV
Status: Recruiting | Type: Observational
Sponsor: German Heart Institute (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other); Deutsche Stiftung für Herzforschung (Other)
Responsible Party: Sponsor
Other Study IDs: mCAV
Record Dates: First submitted 2023-03-13; First posted 2023-04-24 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-07

CONDITIONS: Cardiac Allograft Vasculopathy
Keywords: heart transplantation; cardiac allograft vasculopathy
MeSH Terms: interventions — Echocardiography; Magnetic Resonance Imaging; Magnetocardiography; Shadowing Technique, Histology; Calcium Signaling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- microvascular cardiac allograft vasculopathy: Heart transplant recipients with microvascular cardiac allograft vasculopathy defined by histopathology and invasive index of microvascular resistance.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Magnetic resonance imaging; Diagnostic Test: Magnetocardiography; Diagnostic Test: Histology; Diagnostic Test: Genetics; Diagnostic Test: calcium signaling; Diagnostic Test: IMR; Diagnostic Test: Angio-IMR
- control: Heart transplant recipients without microvascular cardiac allograft vasculopathy defined by histopathology and invasive index of microvascular resistance.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Magnetic resonance imaging; Diagnostic Test: Magnetocardiography; Diagnostic Test: Histology; Diagnostic Test: Genetics; Diagnostic Test: calcium signaling; Diagnostic Test: IMR; Diagnostic Test: Angio-IMR

INTERVENTIONS:
Diagnostic Test: Echocardiography — Echocardiography with afterload change
Diagnostic Test: Magnetic resonance imaging — Stress-MRI
Diagnostic Test: Magnetocardiography — Magnetocardiography
Diagnostic Test: Histology — Histological analysis
Diagnostic Test: Genetics — miRNA sequencing
Diagnostic Test: calcium signaling — cardiomyocyte calcium signaling
Diagnostic Test: IMR — Index of microvascular resistance measurement
Diagnostic Test: Angio-IMR — Angiography derived post-processing index if microvascular resistance

SUMMARY:
The aim of the mCAV study is a comprehensive characterization of the genetic, morphological and functional phenotype of isolated microvascular graft vasculopathy (mCAV) after orthotopic heart transplantation (OHT).

The utilized methods include dynamic echocardiography, magnetic resonance imaging, invasive microvascular resistance measurements, histology, cellular calcium-signaling and magnetocardiography as well as molecular genetic expression analysis (miRNA based).

ELIGIBILITY:
Inclusion Criteria:

* able to consent
* Written consent of the participant after clarification and sufficient time to think about participation
* heart transplant recipient
* Indication for routine invasive diagnostics or due to symptoms
* Exercise tolerant in everyday life - cycling, climbing stairs at least 2 floors at a moderate speed without symptoms of exertion or dyspnea

Exclusion Criteria:

* Addiction or other diseases that do not allow the patient to assess the nature and scope as well as possible consequences of the study
* Patients or their legal guardians who do not sign the declaration of consent or who cannot fully understand it due to a lack of German language skills
* Pregnant women, breastfeeding women
* Severe comorbidities affecting the miRNA profile: diabetes mellitus, malignancy, end-stage renal disease with renal replacement therapy
* Contraindication to the stress test: signs of cardiac decompensation, angina pectoris, dyspnea, hyperthyroidism, GFR <30 ml/min, peripheral arterial disease, pheochromocytoma, angle-closure glaucoma, prostate adenoma, paroxysmal tachycardia, tachycardia atrial fibrillation
* Evidence of an acute rejection or local wall motion disturbances in the resting echocardiography

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Heart transplant recipients
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
mCAV status influences pw-doppler wall motion analysis in echocardiography | at study inclusion
  pw-doppler wall motion analysis is measured with afterload increase
mCAV status influences global longitudinal strain in echocardiography | at study inclusion
  global longitudinal strain is measured by speckle tracking analysis with afterload increase
mCAV status influences diastolic strain in echocardiography | at study inclusion
  diastolic strain is measured by speckle tracking analysis with afterload increase
mCAV status influences cardiac deformity | at study inclusion
  cardiac deformity analysis are performed by MRI
mCAV status influences grade of fibrosis | at study inclusion
  fibrosis grades are measured by MRI
mCAV status influences extracellular volume | at study inclusion
  extracellular volume is measured by MRI
mCAV status influences the circulating miRNA profile | at study inclusion
  circulating miRNA profile is measured by miRNAseq

SECONDARY OUTCOMES:
mCAV status influences the intrinsic cardiac magnetic field | at study inclusion
  the intrinsic cardiac magnetic field is measured by magnetocardiography
mCAV status influences the cellular calcium signaling | at study inclusion
  the cellular calcium is visualized by confocal laser microscopy using electrical stimulation
mCAV status influences subcellular structures | at study inclusion
  mitochondria, T-tubuli are described after visualization by confocal laser microscopy

CONTACTS AND LOCATIONS:
Locations (1):
- DHZC Deutsches Herzzentrum der Charité, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No